CLINICAL TRIAL: NCT04743024
Title: TREAT Child Alcohol Use Disorder (C-AUD) in Eastern Uganda: Screening, Diagnostics, Risk Factors and Handling of Children Drinking Alcohol
Brief Title: TREAT Child Alcohol Use Disorder (C-AUD) in Eastern Uganda
Acronym: TREAT C-AUD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bergen (Other)
Collaborators: The Research Council of Norway (Other); Makerere University (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: RCN project no 285489
Record Dates: First submitted 2020-11-11; First posted 2021-02-08 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Alcohol Abuse; Alcohol Drinking; Alcoholism; Alcohol Use Disorder; Alcohol Dependence; Child Abuse; Child Malnutrition; Child Neglect; Child Mental Disorder; Child, Only
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Child Nutrition Disorders; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine from 3594 children 3594 carer-child pairs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Household: Household carer-child pairs will be included according to age and consent criteria

SUMMARY:
The investigators will investigate the existence of alcohol drinking among children living under adult supervision and care, living within the communities. The investigators will focus on the age group 6-13 years overlapping with the recommended age for primary school attendance. The project is approaching the research topic using quantitative and qualitative methods. The TREAT C-AUD research project will therefore document to which degree alcohol drinking is a problem among children in Mbale, Eastern Uganda.

DETAILED DESCRIPTION:
Uganda has as many other sub-Saharan countries high alcohol consumption per capita and traditions for home brewing. The TREAT C-AUD research project, with partners from Makerere University in Uganda, University of Bergen and Norwegian University of Science and Technology in Norway, will investigate the existence of alcohol drinking among children living under adult supervision and care, living within the communities. The investigators will focus on the age group 6-13 years overlapping with the recommended age for primary school attendance. The project is approaching the research topic from comprehensive perspectives including a large cross-sectional study, interviews with parents and carers, children and stakeholders in the communities, schools and in the health system. The investigators have been including community representatives, expert groups, user groups and stakeholders in the development of screening tools and will do so in interpreting and disseminating the results. The investigators have to take the Covid-19 situation into account both with regard to its effect on the research question at stake and the methods used. The TREAT C-AUD research project will therefore document to which degree alcohol drinking is a problem among children in the communities in Mbale District, Eastern Ugandan. The data collection is capturing cofactors such as other substance use, mental health, parenting, trauma, nutrition and growth. The development of alcohol assessment tools can be used by the health- and school-system for detection and handling of children having problems with alcohol. The investigators will collaborate closely with services in case of identification of children suffering severe harm and adhere to Good Clinical Practice guidelines for ethical conduct, the consent procedure, follow-up and referral.

ELIGIBILITY:
Inclusion Criteria:

Care-giver- child pairs

* Children 6-13 years
* Caregiver of eligible child
* Caregiver adult capable of giving informed consent
* Living in household for minimum 6 months together

Exclusion Criteria:

• Caregiver or child not living in household

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Child-carer
Sampling Method: Probability Sample
Enrollment: 7188 (Estimated)
Dates: Start 2020-12-27 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of alcohol use disorder using context adapted CRAFFT screening tool | 2020-2021
  Period

SECONDARY OUTCOMES:
Parenting: Alabama Parenting questionnaire short form (APQ - 15) | 2020-2021
  The short form includes 15 items scored 0 (never), 1 (almost never), 2 (sometimes), 3 (often), 4 (always) on the five subscales as follows: Involvement (3 qs), Positive Parenting (3 qs), Poor Monitoring/Supervision (3 qs), Inconsistent Discipline (3 qs), Corporal Punishment (3 qs), respectively. No reverse coding necessary when sub-scales reported separately.
Parenting: Conflict Tactic Scale (Original: Straus, 1979, we use: Murray 1995) Version: PARENT-CHILD CONFLICT TACTICS SCALES, FORM CTSPC-CA | 2020-2021
  Parent score: 0=no, 1=yes Parent form: Min= 0, max= 22 High score indicates high level of conflict and violence.
  Child score:
  0 = it has not happened in the past year
  1. = less than monthly
  2. = monthly
  3. = weekly
  4. =daily
  Included subscales:
  Psychological aggression (5 qs), severe assault (4 qs), and very severe assault (4 qs), problems with taking care of child (5 qs) Child form: Min = 0, max = 88 High score indicates high level of conflict and violence.
Child trauma: Child and Adolescent Trauma Screen (CATS) | 2020-2021
  Scored yes (1) or no (0). 16 questions, yes/no Min: 0 Max: 16 The total score is calculated by adding together the score for each of the items where a higher score indicates more traumatic events.
Adult trauma: Stressful Life Events Screening Questionnaire (SLESQ) | 2020-2021
  Scored yes (1) or no (0). 14 questions Min: 0 Max 14 The total score is calculated by adding together the score for each of the items where a higher score indicates more stressful live events.
Post traumatic stress disease (PTSD) 2-item checklist | 2020-2021
  2 questions on clinical and psychological symptoms recorded as: 0=Not at all
  1. A little bit
  2. Moderately
  3. Quite a Bit
  4. Extremely Min-Max: 0-8 A higher score means higher symptom load.
Child mental health: Pediatric symptom checklist (PSC) - child and adolescent version 35 Mental health measures using Pediatric symptom checklist | 2020-2021
  PSC (Pediatric symptom checklist) 35 questions. It is scored from 2 (often), 1 (sometimes), to 0 (never).
  Minimum score= 0, maximum score = 70 The total score is calculated by adding together the score for each of the items where a higher score indicates more impairment.
Carer mental health: Self Reporting questionnaire (SRQ) Mental health measures using Pediatric symptom checklist - child version | 2020-2021
  20 questions. Scored yes (1) or no (0). The total score is calculated by adding together the score for each of the items where a higher score indicates more symptoms of mental illness.
  Min: 0, max: 20
Carer substance use: The alcohol use disorder identification test (AUDIT) | 2020-2021
  10 questions, most reported as increasing frequency. The higher score the more vulnerability to having an alcohol drinking problem.
  Min: 0, max: 20
Dietary diversity- 24 hour recall, food categories as specified by food and agriculture organization 2010 (ISBN 978-92-5-106749-9) | 2020-2021
  A higher score means higher diversity
Food frequency questionnaire | 2020-2021
  the most common food items captured as: 0 = No/never,
  1. = Yes, less than weekly
  2. = 1-3 times/week
  3. = 4-6 time/week
  4. = daily A higher score means a richer, more diversified diet
Household food security-HIFAS | 2020-2021
  6 questions on food security recorded as: 0 = No/never
  1. = Seldom/rare: less than once per month
  2. = Sometimes: 1-2 days last month
  3. = Often: 3-10 days/month
  4. = Very often/usually: more than 10 days last month A higher score means higher household food insecurity.

OTHER OUTCOMES:
Other substance use - sections from Global School Based Health surveys | 2020-2021
  Not a scale, individual questions measuring frequency and number of units used, measured in days per month and units per month.
Height, in cm, 0.1 nearest cm | 2020-2021
  Continuous
Weight, in kg, 0.1 nearest kg | 2020-21
  Continuous
Mid upper arm circumference, cm 0.1 nearest cm | 2020-21
  Continuous
Urine Etg | 2020-21
  Contionuous
Standard U-stix: U-blood, protein, glucose, ketones, nitritt, leukocytes, Ph | 2020-21
  Qualitative reading, positive or negative

CONTACTS AND LOCATIONS:
Overall Officials: Guri Rørtveit, PhD, Study Chair — Leader
Locations (1):
- School of Public Health, Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided
Depending on consent for sharing by study participants

REFERENCES:
- [Result] Engebretsen IMS, Nalugya JS, Skylstad V, Ndeezi G, Akol A, Babirye JN, Nankabirwa V, Tumwine JK. "I feel good when I drink"-detecting childhood-onset alcohol abuse and dependence in a Ugandan community trial cohort. Child Adolesc Psychiatry Ment Health. 2020 Oct 24;14:42. doi: 10.1186/s13034-020-00349-z. eCollection 2020. PMID 33110445
- [Result] Akol A, Makumbi F, Babirye JN, Nalugya JS, Nshemereirwe S, Engebretsen IMS. Does mhGAP training of primary health care providers improve the identification of child- and adolescent mental, neurological or substance use disorders? Results from a randomized controlled trial in Uganda. Glob Ment Health (Camb). 2018 Sep 10;5:e29. doi: 10.1017/gmh.2018.18. eCollection 2018. PMID 30455964
- [Result] Akol A, Nalugya J, Nshemereirwe S, Babirye JN, Engebretsen IMS. Does child and adolescent mental health in-service training result in equivalent knowledge gain among cadres of non-specialist health workers in Uganda? A pre-test post-test study. Int J Ment Health Syst. 2017 Aug 24;11:50. doi: 10.1186/s13033-017-0158-y. eCollection 2017. PMID 28855962
- [Derived] Skylstad V, Aber H, Bakken V, Dierkes J, Iversen SA, Kisaakye E, Kuhl MJ, Nalugya JS, Rayamajhi D, Sebuwufu D, Skar AS, Skokauskas N, Valeckaite N, Wamani H, S Engebretsen IM, Babirye JN; TREAT C-AUD consortium. Child alcohol use disorder in Eastern Uganda: screening, diagnostics, risk factors and management of children drinking alcohol in Uganda (TREAT C-AUD): a mixed-methods research protocol. BMJ Paediatr Open. 2021 Jul 28;5(1):e001214. doi: 10.1136/bmjpo-2021-001214. eCollection 2021. PMID 34345718
- See also: University home page — https://www.uib.no/en/rg/gmh/134660/treat-c-aud-project-page
- Available data/document: Study Protocol: 285489 — https://www.uib.no/en/rg/gmh/134660/treat-c-aud-project-page — IPD will be shared on reasonable request and the official DMP is archived with NFR